CLINICAL TRIAL: NCT02634697
Title: Impact of the Relaxation Response Resiliency Program on Patients With Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Benson-Henry Institute for Mind Body Medicine (Other)
Responsible Party: Principal Investigator, Jeremy n. Ruskin, MD, Director, Cardiac Arrhythmia Service, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015P000552
Record Dates: First submitted 2015-12-10; First posted 2015-12-18 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation; Stress; Quality of Life; Anxiety; Depression; Hostility
Keywords: Atrial Fibrillation; Relaxation Response Resiliency Program Intervention; AF Symptom Severity and Burden; Stress, Anxiety, Depression and Hostility; Quality of Life; AF; QOL; 3RP
MeSH Terms: conditions — Atrial Fibrillation; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3RP Intervention Group (Experimental): AF Patients will undergo the 3RP intervention which will comprise of the following:
  i. One-one-one session: each subject will spend an hour with a clinician to set specific goals for the intervention. They will also answer questionnaires.
  ii. ECG monitoring: Enrolled subjects may be monitored with an ECG at some point after the time of consent up to the day of the one-on-one session, and again after completing the 8 weeks.
  iii. Weeks 1 - 8: subjects will meet with the clinician/staff member as a group once a week for 1.5 hours each where they will be taught a variety of techniques to elicit the relaxation response as well as other cognitive skills.
  At the end of the 4th (mid-point) and 8th (last) weekly session, subjects will answer questionnaires.
  iv. 6 month follow up: 3 months after the final 3RP session to answer questionnaires.
  v. Subjects will be asked to keep track of their AF episodes during the course of the study.
  Interventions: Behavioral: Relaxation Response Resiliency Program
- 3RP Waitlist Control Group (Active Comparator): The Control Group will wait for 6 months (from the time the Intervention group starts the 3RP intervention) and then will undergo the same study procedures as the intervention group - except for the 6 month follow up.
  Interventions: Behavioral: Relaxation Response Resiliency Program

INTERVENTIONS:
Behavioral: Relaxation Response Resiliency Program — 8-week group intervention teaching relaxation and psychological resiliency enhancing skills. Topics include the relaxation response, meditation, and yoga
  Other Names: 3RP

SUMMARY:
The purpose of this study is to determine if an eight week multimodal Relaxation Response Resiliency Program (3RP) intervention can effectively improve symptom severity, frequency and quality of life (Q.O.L) in atrial fibrillation (AF) patients. This will be measured by a reduction in AF symptom score, perceived stress, anxiety, hostility and depression.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a very common cardiovascular disease. Symptoms include dizziness, palpitations, lightheadedness, shortness of breath, fatigue and exercise intolerance. AF is also associated with a high risk of complications like thrombo-embolism and stroke, heart failure, dementia. The presence and severity of these symptoms and complications adversely affect a patient's health related quality of life. Improvement in quality of life (QOL) is an important measure for evaluating response to treatment in AF patients. Depression and anxiety are significant part of the psychosocial burden faced by approximately one-third of AF patients, and are important components that effect QOL in these patients. In this study the investigators will apply the 3RP (Relaxation Response Resiliency Program - developed at the Benson Henry Institute at Massachusetts General Hospital) intervention among AF patients to assess the reduction in their stress, anxiety and depression levels and the reduction in AF symptom burden and severity.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-90 years
2. Diagnosed with documented recurrent symptomatic paroxysmal atrial fibrillation
3. Currently on stable medical therapy for AF and willing to continue on the same treatment regimen for 8 weeks while participating in the study.
4. No current or prior practice of yoga, meditation, guided imagery or other techniques that elicit relaxation response (RR).
5. Able to provide informed consent and to understand written and spoken English.

Exclusion Criteria:

1. End Stage renal failure or heart failure, severe unstable medical or psychiatric disease
2. Patients deemed unable to complete protocol due to cognitive or other reasons.
3. Patients on psychoactive medications will have eligibility determined by the PI or MD co-investigator on a case-by-case basis, and will be admitted to the study if medication is deemed stable

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01-09 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
AF Symptoms Severity and Burden questionnaire | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  A 19-item measure assessing the severity, burden, and impact of one's atrial fibrillation symptoms.
Measure of Current Status (MOCS-A) | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  The MOCS-A is a 13-item measure assessing participants' current self-perceived status on several skills such as: the ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, and choose appropriate coping responses as needed. Responses are made on a 7-point scale with higher scores reflecting higher life satisfaction.

SECONDARY OUTCOMES:
Visual Analog Stress Scale | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  Measures one's distress, stress, and ability to cope with that stress over the past week on a scale from 0 to 10.
Buss-Perry Hostility Scale | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  A 29-item questionnaire that measures a one's levels of aggression.
Cognitive and Affective Mindfulness Scale (CAMS) | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  Measures the degree to which individuals experience their thoughts and feelings.
Cigna Healthy Eating Scale | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  A 7-item self-report instrument that measures behavioral eating.
FACIT-Spirituality | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  Measures spiritual well-being (sense of meaning in life and the sense of strength in one's faith).
Generalized Anxiety Disorder 7-item (GAD-7) | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  A brief measure for assessing generalized anxiety disorder
The Gratitude Questionnaire (GQ-6) | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  The GQ-6 revised is a 6-item measure that assesses individual differences in the proneness to experience gratitude in daily life. Scores range from 6-42, with a higher score indicating a greater sense of gratitude.
Interpersonal Reactivity Index (IRI) | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  The IRI assesses the cognitive and affective dimensions of empathy.
Life Orientation Test (LOT) Optimism Scale | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  The LOT Optimism Scale measures individual differences in generalized optimism versus pessimism.
Medical Outcomes Study (MOS) Social Support Survey | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  The MOS Social Support Survey measures various dimensions of social support.
Positive and Negative Affect Schedule (PANAS) | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  The PANAS comprises two mood scales, one that measures positive affect and the other which measures negative affect.
Patient Health Questionnaire (PHQ) | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  The PHQ measures symptoms of depression and functional impairment.
Lifestyle Questionnaire | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  Measures physical activity and health behaviors.
Pittsburgh Sleep Quality Index (PSQI) | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  Assesses sleep quality and discriminates between good and poor sleepers.
Perceived Stress Scale (PSS-10) | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  The PSS is a widely used psychological instrument for the measurement of the perception of stress. This 10-itam scale is designed to measure the degree to which situations in one's life are appraised, or considered stressful. The scores range from 0-40, with a higher score indicating higher perceived stress. Items were designed to detect how unpredictable, uncontrollable and overloaded respondents find their lives.
Penn State Worry Questionnaire (PSWQ) | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  Measures the trait (or tendency towards) worry in individuals.
RR Adherence Questionnaire | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  Assesses the number of days a week where participants practiced RR skills.
General Self-Efficacy Scale | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  Measures optimistic self-beliefs to cope with a variety of difficult demands in life.
Fatigue and Distress Analogue Scale | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  Measures one's distress and fatigue over the past week on a scale from 0 to 10.
Smoking Questionnaire | Change between Baseline (week 0), mid-intervention (week 4), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  Measures the prevalence and frequency of an individual's smoking habits.
Medication Use Questionnaire | Change between Baseline (week 0), post-intervention (week 9), and 3-month follow up (week 13 or week 26)
  Patients list their medication name, dosage, and frequency.

OTHER OUTCOMES:
Age, Gender, Race, Ethnicity, Marital Status, Education Status, and Employment Status of Patients with AF | Baseline (week 0)
  This questionnaire asks AF patients to report their age, gender, race, ethnicity, marital status, highest level of education, and current employment status.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy N Ruskin, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States